CLINICAL TRIAL: NCT05234853
Title: A Phase I, Open Label, Multicenter Study to Evaluate the Safety and Efficacy of PUR001 Administered Intravenously in Adult Patients With Advanced Solid Tumors
Brief Title: Safety of PUR001 Monotherapy in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Purinomia Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUR001X1101
Record Dates: First submitted 2021-12-27; First posted 2022-02-10 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Monotherapy classic "3+3" design dose escalation and expansion (Experimental)
  Interventions: Drug: PUR001

INTERVENTIONS:
Drug: PUR001 — Monoclonal antibody

SUMMARY:
This is a Phase I, First-In-Human, open label, dose escalation study to evaluate the safety, tolerability, pharmacokinetics, and preliminary anti-cancer activity of PUR001, an anti-CD39 monoclonal antibody, in adult patients with advanced solid tumors, as monotherapy. A "3+3" design will be used to determine MTD and RP2D. .

DETAILED DESCRIPTION:
This is a Phase I, First-In-Human, open label, dose escalation study to evaluate the safety, tolerability, pharmacokinetics, and preliminary anti-cancer activity of PUR001 in adult patients with advanced solid tumors, as monotherapy.

The primary objective of this study is to determine the dose-limiting toxicity(ies) (DLT) and/or maximum tolerated dose (MTD) of PUR001 monotherapy in patients with advanced/metastatic solid tumors.

Study consists of two parts:

Dose Escalation Cohort and Dose Expansion Cohort.

Dose limiting toxicity (DLT) will be evaluated and managed per the pre-defined DLT criteria and rules specified in the protocol. MTD and/or RP2D will be confirmed in a dose confirmation cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Able to sign informed consent and comply with the protocol
2. ≥ 18 years of age, at the time of signing informed consent
3. Histologically or cytologically documented advanced/metastatic solid tumors who have received at least one line of prior systemic chemotherapy and progressed
4. At least one measurable lesion as defined by RECIST V1.1 criteria for solid tumors
5. ECOG performance status of 0 or 1
6. Adequate organ function confirmed at screening and within 10 days of initiating treatment, as evidenced by:

   * Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L
   * Hemoglobin (Hgb) ≥ 8 g/dl
   * Platelets (plt) ≥ 75 × 10^9/L
   * AST/SGOT and ALT/SGPT ≤ 2.5 × Upper Limit of Normal (ULN) or ≤ 5.0 × ULN if liver metastases are present
   * Total bilirubin ≤ 1.5 × ULN
   * Serum creatinine ≤ 1.5 × ULN or calculated creatinine clearance ≥ 30 mL/min (Cockcroft Gault formula
7. Negative pregnancy test within 72 hours before starting study treatment in all pre-menopausal women and women < 12 months after the onset of menopause
8. Must agree to take sufficient contraceptive methods to avoid pregnancy (including male and female participants) during the study and until at least 6 months after ceasing study treatment

Exclusion Criteria:

1. Women who are pregnant or lactating
2. Women of child-bearing potential (WOCBP) who do not use adequate birth control.
3. Patients with untreated brain or central nervous system (CNS) metastases or brain/CNS metastases that have progressed (e.g., evidence of new or enlarging brain metastasis or new neurological symptoms attributable to brain/CNS metastases) Note: Patients with treated brain metastases that are off corticosteroids and have been clinically stable for 28 days are eligible for enrollment
4. Patients with a known concurrent malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, carcinoma in situ of the cervix or other noninvasive or indolent malignancy that has previously undergone potentially curative therapy
5. Impaired cardiac function or significant diseases, including but not limited to any of the following:

   * LVEF < 45% as determined by MUGA scan or ECHO
   * Congenital long QT syndrome
   * QTcF ≥ 480 msec on screening ECG
   * Unstable angina pectoris ≤ 3 months prior to starting study drug
   * Acute myocardial infarction ≤ 3 months prior to starting study drug
6. Patients with uncontrolled hypertension (defined as blood pressure of ≥ 150 mmHg systolic and/or ≥ 90 mmHg diastolic at Screening)
7. Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g., uncontrolled hypertriglyceridemia [triglycerides > 500 mg/dL], or active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with the protocol
8. Patients who have received chemotherapy, targeted therapy, or immunotherapy ≤ 5 half-lives or 3 weeks, whichever is shorter, (except for: 4 weeks for other anti-CD39 monoclonal antibody, 6 weeks for nitrosourea or mitomycin-C) prior to starting study drug
9. Patients who have received wide field radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study drug or who have not recovered from adverse events of prior therapy
10. Patients who have undergone major surgery ≤ 4 weeks prior to starting study drug or who have not recovered from adverse events of prior therapy
11. Patients who are currently receiving treatment with therapeutic doses of warfarin sodium (Coumadin®) or any other coumarin-derivative anticoagulants
12. Known diagnosis of human immunodeficiency virus (HIV) infection (HIV testing is not mandatory; patients with well controlled HIV might be enrolled per investigator's discretion and Sponsor approval).
13. Evidence of active infection with Hepatitis B or Hepatitis C that is not adequately controlled. (For patients with known prior history of Hepatitis B or Hepatitis C, enrollment may be allowed per investigator's discretion and Sponsor approval.)
14. Has a history or current evidence of any condition, therapy, or laboratory abnormality that, in the opinion of the investigator, might confound the results of the trial, interfere with the patient's safe participation and compliance in the trial. For example, conditions that depend on the establishment of collateral circulation, such as peripheral arterial vascular disease, myocardial infraction recovery period, etc.
15. Patients with a clinical history of ≥ grade 3 hypersensitivity reaction (HSR) to biologicals that cannot be controlled by steroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2022-04-28 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) and Maximum Tolerated Dose (MTD), if reached | 1-1.5 years
  Safety and tolerability of PUR001 as a single agent

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events (AEs) | 1-1.5 years
  Safety and tolerability of PUR001 as a single agent. AEs will be assessed per CTCAE v5.0 and may include, but is not limited to, clinically abnormal laboratory tests, physical exams, vital signs, electrocardiograms, and ECOG performance status.
Number of participants with positive Anti-therapeutic antibody (ATA) | 1-1.5 years
  Safety and tolerability of PUR001 as a single agent
Area under the concentration time curve (AUC 0-last) | 1-1.5 years
  Pharmacokinetic (PK) profile of PUR001 as a single agent
Maximum plasma concentration (Cmax) | 1-1.5 years
  Pharmacokinetic (PK) profile of PUR001 as a single agent
Time to Maximum Plasma Concentration (Tmax) | 1-1.5 years
  Pharmacokinetic (PK) profile of PUR001 as a single agent
Half-life (T1/2) | 1-1.5 years
  Pharmacokinetic (PK) profile of PUR001 as a single agent
Mean Residence Time (MRT) | 1-1.5 years
  Pharmacokinetic (PK) profile of PUR001 as a single agent
Volume of Distribution (Vd) | 1-1.5 years
  Pharmacokinetic (PK) profile of PUR001 as a single agent
Objective Response Rate (ORR) | 1-1.5 years
  Preliminary efficacy profile of PUR001 as a single agent
Disease Control Rate (DCR) | 1-1.5 years
  Preliminary efficacy profile of PUR001 as a single agent
Duration of Response (DOR) | 1-1.5 years
  Preliminary efficacy profile of PUR001 as a single agent
Progression free survival (PFS) | 1-1.5 years
  Preliminary efficacy profile of PUR001 as a single agent

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Director — Purinomia Biotech, Inc.
Locations (1):
- The University of Texas MD Anderson Cancer Center, Houston, Texas, United States